CLINICAL TRIAL: NCT06366516
Title: Clinical Validation of ASTN1, DLX1, ITGA4, RXFP3, SOX17, ZNF671 Methylation in HPV Positive Women: a Multi-center RCT From China
Brief Title: Role of Methylation Test Triage in HPV Positive Women
Acronym: MTTRIHPW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Collaborators: Peking Union Medical College Hospital (Other); Chengdu Women's and Children's Central Hospital (Other); Guangdong Women and Children Hospital (Other); Second Hospital of Jilin University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Third Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FUOBGY2024-23
Record Dates: First submitted 2024-03-27; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Precancerous Cervical Lesion
Keywords: Human papillomavirus; High-grade squamous intraepithelial lesion; Methylation; Cervical cancer screening; Triage; Adenocarcinoma in Situ; Cytology
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Adenocarcinoma in Situ | interventions — Colposcopy; Biopsy

STUDY DESIGN:
Intervention Model Description: Women who aged 25 to 65 years are screened for cervical cancer and they are all positive of high-risk HPV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women aged 25-65 years with high-risk HPV infection. (Experimental): Ten thousand women were recruited who aged 25-65 years and they are positive for high-risk HPV.
  Interventions: Diagnostic Test: Methylation Test

INTERVENTIONS:
Diagnostic Test: Methylation Test — Participants who aged 25-65 years with high-risk HPV infection are recruited.To start with,cervical exfoliated cells are collected, coded (according to the actual enrollment sequence), and stored in the pathology department where methylation testing is performed.In addition,patients will underwent colposcopy and biopsy.
  Patients are followed up by cytology, high-risk HPV and methylation tests at 6 and 12 months after enrollment.Cervical conization and hysterectomy will be taken if necessary according to histopathological results. The clinical endpoint is reached when CIN2+ is confirmed by histopathological result.
  Other Names: Liquid-based Cytology Test; High-risk HPV test; Colposcopy; Biopsy

SUMMARY:
The pathological results were used as the gold standard in this study and the investigators analyze the diagnostic value of six gene methylation status (ASTN1 DLX1, ITGA4, RXFP3, SOX17, ZNF671) in triaging high-risk human papillomavirus infection. The sensitivity and specificity of methylation test and cytology in the diagnosis of high-grade cervical lesions are compared in order to providing new methods and basis in improving the accuracy of cervical cancer screening.

DETAILED DESCRIPTION:
The study is divided into two phases, a baseline (cross-sectional) phase and a 1-year follow-up phase. Women who meet the clinical endpoint (i.e. histopathologically confirmed ≥CIN2 after baseline colposcopy/biopsy) are withdrawn from the study. Participants who do not meet the primary endpoint/treat at baseline will invited to participate in the follow-up phase of the trial. Participants included in the follow-up phase are underwent HPV, cytology, and methylation tests at 6 months and 1 year after baseline.Similar to the baseline phase,participants were referred to colposcopy/biopsy if any of the cytology and HPV tests result is positive.

ELIGIBILITY:
Inclusion Criteria:

* aged 25~65 years undergoing cervical cancer screening
* normal for cytology and positive for hrHPV
* informed consent was obtained

Exclusion Criteria:

* pregnant
* with a known history of ablation or treatment with cervical excision within 12 months
* hysterectomy
* chemoradiotherapy
* planning to participate or taking part in another cancer screening, treatment, or vaccination study
* do not meet the inclusion criteria
* give up the trial or naturally dropped out of the follow-up during the observation process
* people who asked to withdraw

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The aim of this study is to evaluate the value of methylation test in high-risk HPV positive women who aged 25 to 65 years for detecting high-grade cervical lesions and cervical cancer.
Enrollment: 10000 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of methylation test in detecting CIN2+. | From date of enrollment until the date of first documented CIN2+,assessed up to 12 months
  The primary variable of methylation test are as follows:clinical sensitivity, clinical specificity, positive predictive value, negative predictive value, positive likelihood ratio, negative likelihood ratio, positive coincidence rate, and negative coincidence rate.

SECONDARY OUTCOMES:
KAPPA value of methylation test. | From date of enrollment until the date of first documented CIN2+,assessed up to 12 months
  KAPPA value is the secondary variable of methylation test which need to meet statistical criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Long Sui, Professor, Study Chair — Obstetrics & Gynecology Hospital of Fudan University; Lan Zhu, Professor, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected data from participants will be shared，including age of patients, the results of cytological examination/high-risk HPV genotyping/methylation test/histopathological, colposcopy impression, and whether cervical conization or hysterectomy were performed before.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: We will apply for a web address to upload all collected clinical data and trial results. The public can send email or request access to the web if any of them needed. After waiting for the principal investigator's consent, the data would be shared by browsing the website.

REFERENCES:
- [Background] Kremer WW, Steenbergen R, Heideman D, Kenter GG, Meijer C. The use of host cell DNA methylation analysis in the detection and management of women with advanced cervical intraepithelial neoplasia: a review. BJOG. 2021 Feb;128(3):504-514. doi: 10.1111/1471-0528.16395. Epub 2020 Aug 9. PMID 32619334
- [Result] Giorgi Rossi P, Carozzi F, Ronco G, Allia E, Bisanzi S, Gillio-Tos A, De Marco L, Rizzolo R, Gustinucci D, Del Mistro A, Frayle H, Confortini M, Iossa A, Cesarini E, Bulletti S, Passamonti B, Gori S, Toniolo L, Barca A, Bonvicini L, Mancuso P, Venturelli F, Benevolo M; the New Technology for Cervical Cancer 2 Working Group. p16/ki67 and E6/E7 mRNA Accuracy and Prognostic Value in Triaging HPV DNA-Positive Women. J Natl Cancer Inst. 2021 Mar 1;113(3):292-300. doi: 10.1093/jnci/djaa105. PMID 32745170
- [Result] van den Helder R, Steenbergen RDM, van Splunter AP, Mom CH, Tjiong MY, Martin I, Rosier-van Dunne FMF, van der Avoort IAM, Bleeker MCG, van Trommel NE. HPV and DNA Methylation Testing in Urine for Cervical Intraepithelial Neoplasia and Cervical Cancer Detection. Clin Cancer Res. 2022 May 13;28(10):2061-2068. doi: 10.1158/1078-0432.CCR-21-3710. PMID 35266975
- [Result] Dovnik A, Poljak M. The Role of Methylation of Host and/or Human Papillomavirus (HPV) DNA in Management of Cervical Intraepithelial Neoplasia Grade 2 (CIN2) Lesions. Int J Mol Sci. 2023 Mar 30;24(7):6479. doi: 10.3390/ijms24076479. PMID 37047452
- [Result] Mazurec K, Trzeszcz M, Mazurec M, Streb J, Halon A, Jach R. Triage Strategies for Non-16/Non-18 HPV-Positive Women in Primary HPV-Based Cervical Cancer Screening: p16/Ki67 Dual Stain vs. Cytology. Cancers (Basel). 2023 Oct 21;15(20):5095. doi: 10.3390/cancers15205095. PMID 37894462
- [Result] Yang S, Wu Y, Wang S, Xu P, Deng Y, Wang M, Liu K, Tian T, Zhu Y, Li N, Zhou L, Dai Z, Kang H. HPV-related methylation-based reclassification and risk stratification of cervical cancer. Mol Oncol. 2020 Sep;14(9):2124-2141. doi: 10.1002/1878-0261.12709. Epub 2020 Jun 2. PMID 32408396
- [Result] Stoler MH, Baker E, Boyle S, Aslam S, Ridder R, Huh WK, Wright TC Jr. Approaches to triage optimization in HPV primary screening: Extended genotyping and p16/Ki-67 dual-stained cytology-Retrospective insights from ATHENA. Int J Cancer. 2020 May 1;146(9):2599-2607. doi: 10.1002/ijc.32669. Epub 2019 Oct 6. PMID 31490545
- [Result] Wright TC Jr, Stoler MH, Ranger-Moore J, Fang Q, Volkir P, Safaeian M, Ridder R. Clinical validation of p16/Ki-67 dual-stained cytology triage of HPV-positive women: Results from the IMPACT trial. Int J Cancer. 2022 Feb 1;150(3):461-471. doi: 10.1002/ijc.33812. Epub 2021 Sep 25. PMID 34536311